CLINICAL TRIAL: NCT06165120
Title: Preputial Graft Versus Preputial Flap in Treatment of Proximal Hypospadias With Marked Ventral Curvature (a Comparative Study)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Ahmed Mohamed Ahmed Mahmoud, Resident at Pediatric Surgery Departemt at Sohag University Hospitals, Sohag University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Soh-Med-23-10-013MS
Record Dates: First submitted 2023-11-22; First posted 2023-12-11 (Actual); Last update posted 2023-12-11 (Actual); Status verified 2023-12

CONDITIONS: Hypospadias, Penoscrotal
MeSH Terms: conditions — Hypospadias

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group A; Bracka's repair group (Active Comparator): This group will undergo Bracka's repair using preputial graft in treatment of proximal hypospadias with marked ventral curvature
  Interventions: Procedure: Bracka's repair using preputial graft
- group B; STPIF repair group (Active Comparator): This group will undergo STPIF repair using preputial flap in treatment of proximal hypospadias with marked ventral curvature
  Interventions: Procedure: STPIF (Staged Transverse Preputial Island Flap) repair using preputial flap

INTERVENTIONS:
Procedure: Bracka's repair using preputial graft — Staged repair:
  1. Correction of ventral chordee: by degloving of the penile skin, transection of the urethral plate &/or ventral corporotomy through the tunica albuginea. This will be according to the degree of ventral chordee after artificial erection test.
  2. Preputial graft placement: a graft will be designed on the inner layer of the preputial hood, according to the length of the urethra defect. Fixation of the free graft will be performed along the whole defective urethral plate. A compression dressing will be used for the transplanted graft. At the end of the surgery, a urinary catheter will be placed through the ectopic meatus.
  3. Tubularisation of the graft: this stage will be performed 6 months later. The new graft will be tubularised over a catheter. Then a protective layer may be made over the tubularization using a dartos or tunica vaginalis flap. After suturing of the penile skin and dressing of the penis, a urethral catheter would be retained for urinary diversion.
  Arms: group A; Bracka's repair group
Procedure: STPIF (Staged Transverse Preputial Island Flap) repair using preputial flap — Staged repair:
  1. Correction of ventral chordee; by degloving of the penile skin, transection of the urethral plate &/or ventral corporotomy through the tunica albuginea. This will be according to the degree of ventral chordee after artificial erection test.
  2. Preputial flap placement: according to the distance between the ectopic meatus and the glans tip, a transverse rectangular flap will be dissected from the inner layer of the dorsal prepuce. The flap will be placed along the defective urethral plate. Eventually, a silicon indwelling catheter will be placed through the ectopic meatus.
  3. Tubularisation of the flap: this stage procedure would be performed 6 months after the first procedure. Tubularisation of the the preputial flap will be done over a catheter. Byar's flaps may be created and transposed to cover the neourethra. Eventually, the penis will be dressed, and a urethral catheter will be retained for urinary diversion.
  Arms: group B; STPIF repair group

SUMMARY:
Hypospadias is a male congenital anomaly characterized by the abnormally located urethral meatus being displaced along the ventral side of the penis along a line from the tip of glans penis to the perineum.

Hypospadias is one of the most common congenital malformations of the male genitourinary system, with a reported global incidence of 0.6-34.2 per 10,000 live births. There is more than one classification for hypospadias. Most commonly, hypospadias is classified into proximal & distal hypospadias which mainly affects the decision for the corrective procedure.

Correction of proximal hypospadias remains a surgical challenge, which is mainly due to the pathological features of proximal hypospadias including a more proximal meatus, severe ventral chordee, and the need to transect the urethral plate during the operation.

The use of a 2-stage repair was found to achieve more satisfactory functional and cosmetic outcomes for proximal hypospadias with severe ventral chordee . Bracka repair, first described in 1995 by Bracka, is a 2-stage repair which uses grafts. This procedure has been improved over time, and recently it has been associated with satisfactory outcomes in proximal hypospadias with severe ventral curvature. Staged transverse preputial island flap urethroplasty (STPIF), first reported by Chen et al., is another 2-stage repair using flaps based on the traditional transverse preputial island flap (TPIF). STPIF has been shown to reduce the difficulty of surgery and the complication rate in management of proximal hypospadias. Thus, both Bracka repair and STPIF are valuable 2-stage methods, and both have achieved promising results. However, there are no available clear comparative data for determination which method has a better outcome and less complications in treating proximal hypospadias.

This study compares Bracka's procedure using preputial grafts and STPIF (Staged Preutial Island Flap) procedure using preputial flaps in surgical correction of proximal hypospadias with marked ventral curvtaure.

ELIGIBILITY:
Inclusion Criteria:

* All patients with proximal hypospadias with marked ventral curvature (>30 degrees) who presented to the outpatient clinic of Department of Pediatric Surgery in Sohag University Hospital.

Exclusion Criteria:

* Patients with insufficient follow up data or those who are non-compliant on follow up.
* Previously circumcised patients.
* Patients with complex urogenital malformations or DSD.
* Patients with ventral curvature less than 30 degrees.
* Patients with crippled hypospadias.

Ages: 6 Months to 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of residual ventral curvature | 1 year
  measured in degrees; if less than 15 degrees it's acceptable, if more than 15 degrees it will need further correction
Incidence of meatal stenosis | 1 year
  calibrated by urethral Hegar's dilators according to the age
Incidence of urethral stricture | 1 year
  calibrated by urethral Hegar's dilators according to the age
Incidence of glans dehiscence | 1 year
  evaluated subjectively by the patients or the parents using questionnaires and objectively by the surgeons
Incidence of urethro-cutaneous fistula | 1 year
  measured in millimeters; if less than 3 millimeters it's a micro-fistula, if it's more than 3 millimeters it's a macro-fistula
Incidence of urethral diverticula formation | 1 year
  evaluated by voiding problems
Incidence of graft/flap fibrosis after the first stage | 1 year
  evaluated objectively by signs of inflammation, necrosis and fibrosis
Percentage of patients with accepted cosmetic appearance | 1 year
  assessed by questionnaires obtained from the patients and/or the parents

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University Hospitals, Sohag, Egypt